CLINICAL TRIAL: NCT03358394
Title: Mindfulness-based Arabic Guided Self-help for Parents of Children With Type 1 Diabetes: A Randomised Pilot Trial.
Brief Title: Mindfulness-based Arabic Guided Self-help for Parents of Children With Type 1 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SHAHAH ALTAMMAR (Other)
Responsible Party: Sponsor-Investigator, SHAHAH ALTAMMAR, PhD Student, University of Sheffield
Organization: University of Sheffield (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Reference Number 016511
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-12

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be asked to complete the outcomes measures anxiety, depression and mindfulness questionnaires at baseline, a week before the start of the intervention and at the end of the intervention time period(i.e., after five weeks).
  Interventions: Behavioral: A human-interventional study
- Control group (Experimental): The control group will be asked to complete the outcomes measures anxiety, depression and mindfulness questionnaires at baseline, a week before the start of the intervention and at the end of the intervention after six weeks.
  At the end of the pilot trial, control group will receive the full intervention. They would be sent the materials week by week as same as the intervention group.
  Interventions: Behavioral: A human-interventional study

INTERVENTIONS:
Behavioral: A human-interventional study — The intervention was developed by Ahmed et al. (2017) and was adapted by the investigators for parents of children with T1D. The researcher has received permission form the author to use the script but, not the audio recordings. As a result, we contacted Saab et al. (2016) to get the permission to use the Arabic audio recording of Mindfulness exercises (i.e., introduction to mindfulness practice and mindfulness breathing).
  The mindfulness script to be used in the current study is based on MBPT. In this study, we will be using the MBPT programme, but tailored to the needs of parents of children with T1D. One of the main changes in our study is that it will be delivered via the Internet. Participants in the original MBPT programme attended in-person sessions however, Rayan et al. (2016) delivered only the first two sessions in person and the rest via telephone

SUMMARY:
Kuwait ranks as the third country worldwide for the incidence of type 1 diabetes (T1D) with an incidence of 37.10 per 100,000 children. A systematic review revealed that anxiety and depression are common in parents of children with T1D . Despite the high incidence rate, only one study to date has examined the psychological impact of diabetes on parents of children with T1D in Kuwait. It was found that 50.8% of parents had elevated levels of anxiety and 46.7% had elevated levels of depression.

Recent research shows that mindfulness is associated with a range of positive outcomes as well as decreased psychological and emotional distress. The earlier A doctor of philosophy (PhD) study found that mindfulness explained large amount of variance in anxiety and depression in a sample of parents of children with T1D. Mindfulness is defined as "paying attention in a particular way, on purpose, in the present moment, and non-judgmentally". The model of mindful parenting can be taught and provided as an intervention to improve psychological outcomes in parents of children with long term health conditions.

In line with this idea, one study examined the effectiveness of a mindfulness-based intervention on perceived stress and psychological anxiety among parents of children with autism spectrum disorder (ASD) in Jordan. The results indicated a significant decrease in stress and psychological distress in the intervention group compared to the comparison group. In the present pilot study, we will extend this work by evaluating a guided self-help a mindfulness intervention that aims to increase mindfulness and reduce psychological distress in parents of children with T1D in Kuwait.

DETAILED DESCRIPTION:
Aims and objectives

The overall aim of this pilot study is to assess the feasibility and acceptability, as well as examine potential effectiveness (from baseline to the end of the intervention), of a self-help online mindfulness-based intervention for Arab parents of children with T1D.

The specific objectives are to:

1. Assess the acceptability of a guided self-help intervention for Arab parents of children with T1D.
2. Ensure recruitment, randomisation and intervention procedures are feasible.
3. Assess time to complete the intervention, for example whether it is feasible for parents to practice mindfulness (10-20 mins) and answer the log sheet daily.
4. Evaluate the ability of the proposed outcome measures (anxiety, depression and mindfulness) to identify change when comparing the mindfulness group to the wait-list control group.

Hypotheses

1. Mindfulness self-help intervention will be an acceptable intervention for parents of children with T1D.
2. The procedures of the pilot study will be feasible (i.e., recruitment, randomisation and deliver of the intervention).
3. The time for practice of mindfulness and completion of the log sheet daily will be feasible.
4. The mindfulness self-help intervention will reduce levels of psychological distress and improve trait mindfulness in some participants.

Participants Sample size of 12-15 per group is recommended for a pilot phase II trial. The investigators need to recruit 30 parents (15 per group) for the pilot trial, which represents approximately half of the potential participants from the pre-existing list (although the investigators hope to recruit up to 40 to allow for some attrition at follow-up). Given that the participants on this list have already taken part in a research study on this topic and have indicated that they would be interested in participating in further studies, the investigators believe that the required recruitment rate is achievable.

Nonetheless, if sufficient participants aren't recruited through pre-existing list the investigators will place a post via Kuwait Diabetes Society on Twitter and Instagram. The post will contain the invitation and the link to the survey.

Randomization Participants will be randomly assigned to either the mindfulness intervention group or the wait list group using the randomization.com website http://www.randomization.com.

Design. This study will be a randomised pilot trial of a guided self- help online mindfulness intervention for parents of children with T1D. The study will have two independent variables: one between-participant variable with two levels, treatment condition (mindfulness-based guided self-help vs. waiting list group), and one within-participants variable with two levels, time (time one and time two). The dependent variables are anxiety, depression and mindfulness.

In the current study, the mindfulness guided self-help intervention will be delivered over a five-week period. The mindfulness training's are MP3 ( i.e., is an audio coding format for digital audio) self-help audio recordings that will be delivered online (i.e., Mindfulness introduction, Mindful breathing). A Clinical Psychologist, Hend Saab, recorded these audios files. Other mindfulness skills will be provided to the parents as a script (PDF file), for example mindfulness eating. Potential participants asked to read the information sheet and give their consent to participate in the current study.

The first session will be delivered using a pre-recorded video. The pre-recorded video will be initiated by the investigators and sent to all participants in the intervention group at the same day and time. After participants have watched the first pre-recorded video session they will be required to tick a box to indicate that they have watched the introduction. Once they have finished watching the introductory pre-recorded video, this will be followed by a brief description of the five core mindfulness skills and mindfulness breathing guided practice. Week two, involves mindfulness breathing guided practice, mindfulness body scan guided practice and integrates mindfulness into other aspects of life. From the third session till the fifth session, parents will require to practice mindfulness breathing guided practice daily and other assignments using the log sheet.

During the intervention, participants will receive guided support in the form of a weekly 30 minute phone call. The investigators will conduct the guided support phone calls. The guidance will consist of: 10 minutes reviewing previous assignment (i.e., mindfulness breathing exercise) for the last week, 15 minutes introducing, delivering and discussing the next mindfulness exercises, and finally 5 minutes for questions. In order to ensure intervention fidelity, a checklist will be used for each phone call. Participants will also receive supportive emails per week to encourage them to practice. Feedback on the acceptability and feasibility of the intervention materials will also be sought from parents (intervention group) of children with T1D at the end of the intervention.

Data Analyses. Statistical analysis will be carried out with statistical package for the social sciences (SPSS). Descriptive analysis (i.e., frequencies, means and standard deviations) will be calculated for all demographics and clinical variables. Descriptive results will include recruitment numbers, completions, dropout rates, and missing data. In addition, mean scores will be calculated for the participants' rating of the intervention's acceptability and frequency. Changes in the three outcome measures in each group from baseline to post-intervention will be assessed by measuring by a series of 2 (group) by 2 (time) ANOVAs.

ELIGIBILITY:
Participants will comprise Kuwaiti parents of children with type 1 diabetes with elevated levels of psychological distress (anxiety or/and depression) who participated in a previous study as part of the PhD research.

Inclusion criteria

Participants included in this study must be:

* Kuwaiti parents of children diagnosed with T1D.
* Children aged 15 and under.
* Have Internet access.
* Arabic speakers.

Exclusion criteria

Participants will be excluded from the study if they are:

• Parents of children diagnosed with type 2 diabetes (T2D).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-02-26 (Estimated); Study Completion 2018-05-16 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder Scale (GAD-7) | 3 minutes
  The GAD-7 is a widely used measure to assess anxiety; seven items have excellent reliability (α = .92) and validity. Items are rated at 4-point scales to produce a total score that can range from 0 to 21.GAD has been translated into Arabic
The Patient Health Questionnaire (PHQ-9). | 3 minutes
  The PHQ-9 has a good reliability (α= .89). It is based on the diagnostic and statistical manual of mental disorders (DSM-IV) criteria for depression disorder. The measure contains 9 items rated on 4-point response scales. Scores can range from 0 to 27. PHQ has been translated into Arabic.
Mindfulness | 10 minutes
  Trait mindfulness will be measured by the the five-facet mindfulness questionnaire short-form (FFMQ-SF). This has 24 questions, which assess the five facets of mindfulness (observing, describing, acting with awareness, nonjudging and nonreacting). The FFMQ-SF is a reliable and valid measure: observing (α =. 81), describing (α =. 87), acting with awareness (α =. 83), non-judging (α =. 83) and non-reacting (α =. 75). The Mindfulness questionnaire has been translated into Arabic.

CONTACTS AND LOCATIONS:
Overall Officials: SHAHAH M ALTAMMAR, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Shahah Altammar, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnard K, Thomas S, Royle P, Noyes K, Waugh N. Fear of hypoglycaemia in parents of young children with type 1 diabetes: a systematic review. BMC Pediatr. 2010 Jul 15;10:50. doi: 10.1186/1471-2431-10-50. PMID 20633252
- [Background] Al-Tammar, S., Norman, P., & Thompson, A. (2017). The Role of Mindfulness and Illness Pereceptions in Psychological Outcomes in Parents of Children with Diabetes. Paper presented at the 31st Annual Conference of the European Health Psychology Society, Padova, Italy.
- [Background] Brown, K. W., Ryan, R. M., & Creswell, J. D. Addressing fundamental questions about mindfulness. Psychological Inquiry, 18, 272-28, 2007.
- [Background] Hayes, S. C., Follette, V. M., & Linehan, M. M. (2011). Mindfulness and Acceptance: Expanding the Cognitive-Behavioral Tradition: Guilford Publications.
- [Background] Piet J, Wurtzen H, Zachariae R. The effect of mindfulness-based therapy on symptoms of anxiety and depression in adult cancer patients and survivors: a systematic review and meta-analysis. J Consult Clin Psychol. 2012 Dec;80(6):1007-20. doi: 10.1037/a0028329. Epub 2012 May 7. PMID 22563637
- [Background] Kabat-Zinn, J. (1994). Wherever you go, there you are: Mindfulness meditation in everyday life. New York: Hyperion.
- [Background] Bögels, S. M., Hellemans, J., van Deursen, S., Römer, M., & van der Meulen, R. (2014). Mindful parenting in mental health care: effects on parental and child psychopathology, parental stress, parenting, coparenting, and marital functioning. Mindfulness, 5, 536-551. doi:10.1007/s12671-013-0209-7
- [Background] Rayan A, Ahmad M. Effectiveness of mindfulness-based interventions on quality of life and positive reappraisal coping among parents of children with autism spectrum disorder. Res Dev Disabil. 2016 Aug;55:185-96. doi: 10.1016/j.ridd.2016.04.002. Epub 2016 Apr 22. PMID 27107368
- [Background] Hertzog MA. Considerations in determining sample size for pilot studies. Res Nurs Health. 2008 Apr;31(2):180-91. doi: 10.1002/nur.20247. PMID 18183564
- [Background] Julious, S. A. (2005). Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics, 4(4), 287-291. doi:10.1002/pst.185
- [Background] Ferraioli, S. J., & Harris, S. L. (2013). Comparative effects of mindfulness and skills-based parent training programs for parents of children with autism: feasibility and preliminary outcome data. Mindfulness, 4(2), 89-101.
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Bergomi, C., Tschacher, W., & Kupper, Z. (2013). The Assessment of Mindfulness with Self-Report Measures: Existing Scales and Open Issues. Mindfulness, 4(3), 191-202. doi:10.1007/s12671-012-0110-9
- See also: International Diabetes Federation. (2015). IDF Diabetes Atlas. — http://www.diabetesatlas.org